CLINICAL TRIAL: NCT00298402
Title: The Role of Macrophages in the Pathophysiology of Smokers' Lung
Brief Title: Macrophages in Smokers' Lung
Status: Withdrawn | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Other Study IDs: 05/Q0404/87
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis
Keywords: macrophage; MMP; CT scan
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Cigarette smoking causes an increase in inflammation in the lungs. In about 20% of smokers this inflammation leads to damage in lungs including making holes in the lung tissue. This damage can not be repaired and these people find it very difficult to breathe. One of the problems with this disease called chronic obstructive pulmonary disease, or COPD for short, is that by the time patients visit their doctor with symptoms, the damage has already been done. At the moment, there is no way to predict which smokers will go on to develop COPD. The aim of this research is to look at smokers who breathe normally and use an imaging technique called a CT scan, to look at their lungs in more detail. Some of these people will have spots on their scan which may be caused by inflammation. We want to look at the cells at these spots to see if they make more proteins and enzymes that cause lung damage when compared to people that do not have these spots. We would then be able to predict which smokers are likely to develop COPD and treat them early before they have damaged their lungs.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease, or COPD for short, will be 3rd biggest killer in the world by 2020. The major cause of this disease is cigarette smoking, but only about 15-20% of smokers will develop COPD. In this disease, the lung becomes damaged and patients can not breathe properly. This damage can not be repaired therefore at the moment there are no good treatements for COPD. By the time a patient visits their doctor with symptoms the damage is already done. Therefore in this study we want to look at the lungs of smokers that feel well and can breathe normally. We believe that much of the damage to the lung in COPD is caused by inflammation. In particular, there are more inflammatory cells called macrophages in the lungs of these patients. These macrophages normally protect the lung when we inhale particles like dust and are also inportant to fight infections. In COPD, these macrophages are out of control and produce huge amounts of enzymes that break down lung tissue and more proteins that cause inflammation. We want to see if we can find these macrophages in the lungs of smokers before they get COPD. Recently, a 5 and a half year study showed that some smokers that can breathe normally have increased inflammation in their lungs. This can be seen using a scan called a CT scan. On the CT scan, these areas look like spots. When these smokers had another scan 5 and half years later, in some cases these spots had become holes in their lung. This is called emphysema and is one of the characteristics of COPD. We want to know whether the macrophages in these smokers cause this damage. If this is the case, we have two separate findings from this study. Firstly, we could look at macrophages and predict which smokers will develop COPD and secondly, try and develop new treatments to stop the macrophages from producing all proteins that cause inflammation.

ELIGIBILITY:
Inclusion Criteria:

All healthy smoking volunteers in trials will meet the following criteria:

Age 21-70 years. Smoking history of at least 10 pack years. (1 pack year = 20 cigarettes per day for 1 year).

No history of respiratory or allergic disease. Normal baseline spirometry as predicted for age, sex and height. No history of upper respiratory tract infection in the preceding six weeks. Not taking regular medication -

Exclusion Criteria:

Subjects will not included in this study if they meet any of the following exclusion criteria:

Clinically significant findings in the medical history or on physical examination.

Pregnant women or mothers who are breastfeeding. Subjects who are unable to give informed consent -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Athol Wells, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Imperial College London, London, United Kingdom